Project title: Immediate Loading and Fully Guided Surgery: Single Implants

Official title: Immediate loading of single implants, guided surgery and intraoral scanning: a

non-randomized study

NCT04061694

Includes: Statistical analysis plan

Date: 2019-10-08

## Statistical analysis plan

All data were statistically analyzed by one examiner, who did not take part in any of the clinical procedures. The software used was the Statistical Package for the Social Sciences (SPSS) version 25 (SPSS Inc., Chicago, IL). The data were tabulated, and from these measurements mean, standard deviation (SD), minimum and maximum were calculated. Kolmogorov–Smirnov test was performed to evaluate the normal distribution of the variables, and Levene's test evaluated homoscedasticity. The performed tests for two independent groups and two dependent groups were Student's t-test or Mann-Whitney test and Wilcoxon signed-rank test, depending on the normality. Pearson's chi-squared or Fisher's exact test was performed for categorical variables, depending on the expected count of events in a 2×2 contingency table. For DIL, correlation and linear regression were performed to check the relationship between PES, survival and implants position deviations. The degree of statistical significance was considered p < 0.05.